CLINICAL TRIAL: NCT02088411
Title: The Safety and Efficacy of an Enzyme Combination in Managing Knee Osteoarthritis Pain in Adults: a Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: The Safety and Efficacy of an Enzyme Combination in Managing Knee Osteoarthritis Pain in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atrium Innovations (Industry)
Collaborators: Mucos Pharma GmbH, Oberhaching, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MU-699412
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Wobenzym; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac; Wobenzym

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diclofenac (Active Comparator): Subjects assigned to receive 1 tablet of Diclofenac Sodium (50 mg) and two tablets of an indistinguishable placebo three times daily for a duration of 12 weeks.
  Interventions: Drug: Diclofenac
- Wobenzym (Active Comparator): Subjects assigned to receive 2 tablets of Wobenzym(R) and 1 tablet of an indistinguishable placebo three times daily for a duration of 12 weeks.
  Interventions: Dietary Supplement: Wobenzym
- Placebo (Placebo Comparator): Subjects assigned to receive three tablets of an indistinguishable placebo three times daily for a duration of 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac
  Arms: Diclofenac
Dietary Supplement: Wobenzym
  Arms: Wobenzym
Other: Placebo
  Arms: Placebo

SUMMARY:
The aim of this randomized, double-blind, placebo-controlled, comparator-controlled trial was to evaluate the safety and efficacy of an enzyme combination, as Wobenzym®, in adults with moderate-to-severe osteoarthritis (OA) of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis confirmed by radiography or tomography
* Lequesne Functional Index score of 10-14
* WOMAC-A pain subscale score greater than or equal to 25

Exclusion Criteria:

* History of knee trauma
* History of joint infection
* History of joint surgery
* History of intra-articular injection (viscotherapy)
* History of gastrointestinal diseases
* Use of corticosteroids
* Use of COX-II inhibitors
* Use of glucosamine/chondroitin
* Known sensitivity to paracetamol
* Known sensitivity to non-steroidal anti-inflammatory drugs (NSAIDs)
* Known sensitivity to oral enzymes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-11; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

PRIMARY OUTCOMES:
Lequesne Functional Index | Change from baseline to 12 weeks
  Self-assessment of the affected knee joint by physician interview using the Lequesne Functional Index (providing an estimate of the degree of pain associated with the affected joint, the maximum distance talked, and activities of daily living).

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Index version 3.0 subscale for pain (WOMAC-A) | Change from baseline to 12 weeks
Western Ontario and McMaster Universities Index version 3.0 subscale for joint stiffness (WOMAC-B) | Change from baseline to 12 weeks
Western Ontario and McMaster Universities Index version 3.0 subscale for joint function (WOMAC-C) | Change from baseline to 12 weeks
Paracetamol Consumption | Change from baseline to 12 weeks
  Number of paracetamol tablets consumed during the study by subjects
Indices of systemic inflammation | Change from baseline to 12 weeks
  Erythrocyte sedimentation rates at 1 and 2 hours and serum concentration of C-reactive protein
Adverse Events | Through baseline to 12 weeks
  Any complications throughout study.

CONTACTS AND LOCATIONS:
Locations (1):
- Mucos Pharma GmbH & Co, Oberhaching, Germany